CLINICAL TRIAL: NCT04291183
Title: The Effect Of Horticultural Therapy On The Level Of Happiness And Loneliness Of Elderly Living In Nursing Home
Brief Title: Elderly Who Received Horticulturel Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Seda CEVHEROĞLU, PhD Student of Nursing / Senior Instructor Department of Nursing, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IstanbulUC2
Record Dates: First submitted 2020-02-28; First posted 2020-03-02 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Horticultural Therapy; Elderly; Happiness; Loneliness
Keywords: horticultural therapy; elderly; nursing home; happiness; loneliness
MeSH Terms: interventions — Horticultural Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- elderly people to undergo hortic culture therapy (Experimental): Horticultural Therapy will be applied to the elderly in the experimental group in the form of two days a week visit for eight weeks. Flower and vegetable seedlings suitable for the season will be planted in the garden with the elderly. The elderly will be asked to take care of the plants they planted every day (irrigation and collecting extra herbs) and the elderly people will be observed by doing these processes twice a week
  Interventions: Behavioral: horticultural therapy
- elderly people who will not receive horticultural therapy (No Intervention): pre-test data forms will be applied to the control group. Post-test data forms will be reapplied after 8 weeks

INTERVENTIONS:
Behavioral: horticultural therapy — Flowers and vegetables will be planted with the elderly. Growth of plants planted with the elderly will be observed and maintained
  Arms: elderly people to undergo hortic culture therapy

SUMMARY:
Horticultural Therapy (HT) method refers to the process of using gardening as a method to maintain and improve the existing health status of the individual, which can be applied by healthcare professionals. Horticultural therapy method is an application that positively contributes to the cognitive, physical, social, emotional processes and entertainment processes of the elderly. Collins and O 'Callaghan (2008 ) and Yao and Chen (2016) showed that older individuals with serious illness and weakness had improved health outcomes when they were busy with plants. In a study by Yao and Chen (2016); Individuals aged 65 years and older were treated with HT once a week for eight weeks, and an increase in daily life activities, happiness and interpersonal affinity was observed. In another semi-experimental study by Tse (2010), elderly individuals were given HT for eight weeks, after which an increase in life satisfaction and social communication of the elderly and a significant decrease in loneliness were found. These results showed that HT can be used for therapeutic purposes in the elderly.

While horticultural therapy is used as a therapeutic approach for the elderly in nursing homes, there is still no such study in the geography we live in. The research was planned to determine the effect of hortic culture therapy on the loneliness and happiness levels of the elderly living in the nursing home.

DETAILED DESCRIPTION:
In recent years, the elderly population is increasing due to the decrease in the fertility rate in our country, the lifetime due to the improvement in health conditions, the prevention of diseases before they occur as a result of the developments in medicine and technology and that they can be treated successfully even if they occur.

In our country, due to rapid population growth, industrialization and urbanization, transformation into a nuclear family due to internal and external migration, the presence of economic problems, women's participation in working life, young people's perspective on old age, intergenerational communication disorders and addiction make the home care of the elderly difficult and the elderly are placed in different institutions from the family environment. The opportunities of the elderly who go to the institution to get to know and adapt to the environment are lost, and the elderly individual may have feelings such as isolation, loneliness and feeling worthless.

The phenomenon of loneliness is seen in all age groups, but it is a problem specific to the elderly. Loneliness is a common and disturbing problem for many elderly people. The emotional support of elderly individuals is not sufficient, and their friendship relationships are limited, which increases their loneliness. Social support systems, elderly caregivers and healthcare professionals play an important role in coping with loneliness problems and high levels of happiness in the nursing home.

Horticultural Therapy (HT) method refers to the process of using gardening as a method to maintain and improve the existing health status of the individual, which can be applied by healthcare professionals. Horticultural therapy method is an application that positively contributes to the cognitive, physical, social, emotional processes and entertainment processes of the elderly. Collins and O 'Callaghan (2008 ) and Yao and Chen (2016) showed that older individuals with serious illness and weakness had improved health outcomes when they were busy with plants. In a study by Yao and Chen (2016); Individuals aged 65 years and older were treated with HT once a week for eight weeks, and an increase in daily life activities, happiness and interpersonal affinity was observed. In another semi-experimental study by Tse (2010), elderly individuals were given HT for eight weeks, after which an increase in life satisfaction and social communication of the elderly and a significant decrease in loneliness were found. These results showed that HT can be used for therapeutic purposes in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Being 65 or older
* Ability to understand and respond to research guidelines
* Ability to act independently
* No known allergic disease.

Exclusion Criteria:

* Having a diagnosed psychiatric disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-03-11 (Estimated); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
The Loneliness Scale for the Elderly. | 6 months
  Applying garden culture treatment for the elderly who stay in the nursing home. It has been developed for use in determining the loneliness level of the elderly. The scale, which has 11 items in total, consists of two sub-dimensions: six items (2, 3, 5, 6, 9, 10) of the scale, negative items that measure emotional loneliness; five items (1, 4, 7, 8, 11) are positive items that measure social loneliness.
  Total loneliness can be divided into four levels: Level 1; not alone / feeling lonely (score 0-4); Level 2; acceptable loneliness (score 5-14); Level 3; very lonely (points 15-18); Level 4; Very intense loneliness (score 19-22). The lowest score to be taken from the scale is 0, the highest score is 22. The Cronbach's alpha of the scale is α = .85.
The Subjective Happiness Scale. | 6 months
  Applying radicultural therapy for the elderly who stay in the nursing home. Subjective Happiness Scale consists of 4 descriptive items. Item 4 of the scale is reversed. Although there are no sub-dimensions of the scale, minimum 4 and maximum 28 points are obtained from the scale. High scores to be obtained from the scale indicate that the subjective happiness of the individual is high.Cronbach α reliability coefficient was found as .86

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Unıversıty- Cerrahpaşa, Istanbul, Istanbul/ Şişli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kamioka H, Tsutani K, Yamada M, Park H, Okuizumi H, Honda T, Okada S, Park SJ, Kitayuguchi J, Abe T, Handa S, Mutoh Y. Effectiveness of horticultural therapy: a systematic review of randomized controlled trials. Complement Ther Med. 2014 Oct;22(5):930-43. doi: 10.1016/j.ctim.2014.08.009. Epub 2014 Sep 1. PMID 25440385
- [Result] Kim KH, Park SA. Horticultural therapy program for middle-aged women's depression, anxiety, and self-identify. Complement Ther Med. 2018 Aug;39:154-159. doi: 10.1016/j.ctim.2018.06.008. Epub 2018 Jun 26. PMID 30012387
- [Result] Ng KST, Sia A, Ng MKW, Tan CTY, Chan HY, Tan CH, Rawtaer I, Feng L, Mahendran R, Larbi A, Kua EH, Ho RCM. Effects of Horticultural Therapy on Asian Older Adults: A Randomized Controlled Trial. Int J Environ Res Public Health. 2018 Aug 9;15(8):1705. doi: 10.3390/ijerph15081705. PMID 30096932
- [Result] Chan HY, Ho RC, Mahendran R, Ng KS, Tam WW, Rawtaer I, Tan CH, Larbi A, Feng L, Sia A, Ng MK, Gan GL, Kua EH. Effects of horticultural therapy on elderly' health: protocol of a randomized controlled trial. BMC Geriatr. 2017 Aug 29;17(1):192. doi: 10.1186/s12877-017-0588-z. PMID 28851276
- [Result] Nicholas SO, Giang AT, Yap PLK. The Effectiveness of Horticultural Therapy on Older Adults: A Systematic Review. J Am Med Dir Assoc. 2019 Oct;20(10):1351.e1-1351.e11. doi: 10.1016/j.jamda.2019.06.021. Epub 2019 Aug 8. PMID 31402135
- [Result] Lo SKL, Lam WYY, Kwan RYC, Tse MMY, Lau JKH, Lai CKY. Effects of horticultural therapy: Perspectives of frail and pre-frail older nursing home residents. Nurs Open. 2019 Jul 3;6(3):1230-1236. doi: 10.1002/nop2.323. eCollection 2019 Jul. PMID 31367449
- [Result] Soderback I, Soderstrom M, Schalander E. Horticultural therapy: the 'healing garden'and gardening in rehabilitation measures at Danderyd Hospital Rehabilitation Clinic, Sweden. Pediatr Rehabil. 2004 Oct-Dec;7(4):245-60. doi: 10.1080/13638490410001711416. PMID 15513768